CLINICAL TRIAL: NCT05493800
Title: A Phase IIa, Multi-center, Dose-finding Study to Evaluate Safety and Efficacy for Prevention of Oral Mucositis and PK of MIT-001 in Patients With Lymphoma or Multiple Myeloma Receiving Conditioning Chemotherapy Followed by Auto HSCT
Brief Title: Evaluate the Safety and Efficacy for Oral Mucositis Prevention of MIT-001 in Auto HSCT
Acronym: Capella
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: MitoImmune Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MIT001-OM-02
Record Dates: First submitted 2022-08-03; First posted 2022-08-09 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Oral Mucositis; Lymphoma; Multiple Myeloma; Hematologic Cancer
Keywords: oral mucositis; MIT-001; auto HSCT; HSCT; hematopoietic stem cell transplantation; ferroptosis inhibitor; necrosis inhibitor
MeSH Terms: conditions — Stomatitis; Lymphoma; Multiple Myeloma; Hematologic Neoplasms | interventions — Saline Solution

STUDY DESIGN:
Intervention Model Description: Part 1 was completed with 16 patients and open label design to to evaluate the pharmacokinetic characteristics, efficacy, and safety of MIT-001 on prevention effect of MIT-001 in combination with conditioning regimen in auto-HSCT. 5mg as low dose and 20mg as high dose of MIT-001 were determined as RP2D through steering comittee and optional group of 30mg was not needed at Part 1 because low level of MIT-001 was enough to show efficacy and safety of MIT-001.
  In Part 2, it's to determine the optimal dose (recommended part 2 dose (RP2D)) of MIT-001 in combination with conditioning regimen in auto-HSCT.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Part I: open label
  Part II: double blind, randomized, and Placebo controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Part 1, MIT-001 5 mg group (Experimental): Part 1, MIT-001 5 mg, once a day IV administration for 30 minutes before conditioning regimen administration 0.5~1 hr.
  5 subject were enrolled sequentially.
  Interventions: Drug: MIT-001
- Part 1, MIT-001 10 mg group (Experimental): Part 1, MIT-001 10 mg, once a day IV administration for 30 minutes before conditioning regimen administration 0.5~1 hr.
  6 subjects were enrolled sequentially.
  Interventions: Drug: MIT-001
- Part 1, MIT-001 20 mg group (Experimental): Part 1, MIT-001 20 mg, once a day IV administration for 30 minutes before conditioning regimen administration 0.5~1 hr.
  5 subjects were enrolled sequentially.
  Interventions: Drug: MIT-001
- Part 1, MIT-001 30 mg group (Experimental): Part 1, MIT-001 30 mg, once a day IV administration for 30 minutes before conditioning regimen administration 0.5~1 hr.
  It was optional but did not ptoceed according to Steering committee's decision because low level of MIT-001 is enough to show the efficacy and safety of MIT-001.
  Interventions: Drug: MIT-001
- Part 2, 5mg of MIT-001 low dose group (Experimental): Part 2, MIT-001 low dose, once a day IV administration for 30 minutes before conditioning regimen administration 0.5~1 hr.
  15 subject will be enrolled parallelly.
  Interventions: Drug: MIT-001
- Part 2, 20mg of MIT-001 high dose group (Experimental): Part 2, MIT-001 high dose, once a day IV administration for 30 minutes before conditioning regimen administration 0.5~1 hr.
  15 subject will be enrolled parallelly.
  Interventions: Drug: MIT-001
- Part 2, placebo(normal saline) group (Placebo Comparator): Part 2, placebo(normal saline), once a day IV administration for 30 minutes before conditioning regimen administration 0.5~1 hr.
  15 subject will be enrolled parallelly.
  Interventions: Drug: normal saline

INTERVENTIONS:
Drug: MIT-001 — Corresponding dose of MIT-001 IV injection during 0.5~1hr
  Arms: Part 1, MIT-001 10 mg group; Part 1, MIT-001 20 mg group; Part 1, MIT-001 30 mg group; Part 1, MIT-001 5 mg group; Part 2, 20mg of MIT-001 high dose group; Part 2, 5mg of MIT-001 low dose group
Drug: normal saline — normal saline IV injection
  Other Names: placebo
  Arms: Part 2, placebo(normal saline) group

SUMMARY:
Evaluate the efficacy and safety for the prevention of oral mucositis and PK of MIT-001 for lymphoma or multiple myeloma patients receiving conditioning chemotherapy for autologous hematopoietic stem cell transplantation(auto-HSCT).

DETAILED DESCRIPTION:
In Part 1, it was to determine Recommended Part 2 Dose(RP2D) the prevention effect of MIT-001 in combination with conditioning regimen in autologous hematopoietic stem cell transplantation(auto-HSCT) and to evaluate the pharmacokinetic characteristics of MIT-001.

In Part 2, it's to determine the optimal dose of MIT-001 in combination with conditioning regimen in auto-HSCT.

This clinical trial consists of a 28-days of screening period, 4 to 9 days of conditioning chemotherapy with MIT-001 treatment, auto-HSCT and a 14-days of follow-up and recovery period.

MIT-001 group consists of 5 mg (group 1), 10 mg (group 2), and 20mg (group 3), and the subject will be assigned to from 5 mg of MIT-001 sequentially.

After completion of MIT-001 administration from all 3 MIT-001 groups, Steering Committee (SC) was convened and reviewed the safety and efficacy to determine one of the followings.

* Determine whether the next dose (Group 4: 30 mg) in Part 1: It was not proceeded.
* Determine the RP2D to enter Part 2 phase: 5mg as low dose, 20mg as high dose for Part 2 The investigators will continuously monitor the safety of MIT-001, and can request the steering committee call at any time, and can be carefully reviewed the data such as safety and efficacy.

In Part 2, the subjects are randomly assigned to either one of MIT-001 treatment groups (high-dose, low-dose among RP2D) and placebo at a ratio of 1: 1: 1. If two or more conditioning regimen are determined, conditioning regimen can be considered the stratification factor. Subject will be randomly assigned to either group in blinded method.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged 19 to 70 years old
2. Patients with lymphoma or multiple myeloma planned for receiving one of the following conditioning chemotherapy followed by autologous hematopoietic stem cell transplantation

   * BuCyE Regimen: Busulfan (iv) 3.2 mg/kg (Day 1, Day 2, Day 3) + Etoposide (iv) 400 mg/m² (Day 3, Day 4) + Cyclophosphamide (iv) 50 mg/kg/Mesna (iv) 50 mg/kg (Day 5, Day 6), and autologous HSCT after 1 day rest after completion of 6 days of conditioning chemotherapy
   * BMT Regimen: Busulfan (iv) 2.4 mg/kg (Day 1, Day 2, Day 3) + Melphalan (iv) 40 mg/m2 (Day 4, Day 5) + Thiotepa (iv) 200 mg/ m2 (Day 6, Day 7), and autologous HSCT after 1 day rest after completion of 7 days of conditioning chemotherapy
   * Melphalan Regimen: Melphalan (iv) 100 mg/m2 (Day 1, Day 2), and autologous HSCT after 1 day rest after completion of 2 days of conditioning chemotherapy
   * BuMel Regimen: Busulfan (iv) 3.2 mg/kg (Day 1, Day 2, Day 3) + Melphalan (iv) 140 mg/m2 (Day 4), and autologous HSCT after 1 day rest after completion of 4 days of conditioning chemotherapy (In part 2, BUCYE, BMT and MELPHALAN regimens are allowed.)
3. Patients who have not received a hematopoietic stem cell transplant before
4. Patients with Body Mass Index (BMI) 35 or less
5. Patients who have prepared at least 2 x 10^6 CD34+ cell/kg
6. Patients whose hematologic, kidney and liver functions were confirmed to be proper through the following laboratory test results last measured within 8 days prior to the investigational product(IP) administration Laboratory endpoint Required limit for inclusion Absolute neutrophil count (ANC) ≥ 1,000/mm^3 Hemoglobin (Hb) ≥ 9.0 g/dL Platelet count ≥ 100,000/mm^3 Total bilirubin (TB) ≤ 2 mg/Dl AST and ALT ≤ 3.0 x ULN(if liver metastasis, ≤ 5 x ULN) Prothrombin time (PT) INR ≤ 1.5 (if taking warfarin, < 3) Serum creatinine or creatinine clearance (CrCl) < 2 mg/dL or≥ 60 mL/min
7. Patients with Eastern Cooperative Oncology Group performance status (ECOG-PS) of 0 or 1
8. Patients who voluntarily decided to participate in this study after being informed of the study information, and provided written consent to faithfully comply with the study requirements

Exclusion Criteria:

1. Patients who has the following medical history or concomitant diseases at screening

   * Patients with oral mucositis or oral ulcer at screening
   * Patients who have severe infections or other uncontrolled active infectious diseases at screening that require administration of antibiotics, antibacterial agents, antifungal agents, antivirals, etc. (e.g., Human Immunodeficiency Virus positive, active hepatitis B or active hepatitis C, etc.) However, in case of administration of antiviral drugs in patients with hepatitis B or C infection, whose disease is controlled, the subjects can be enrolled.
   * Patients who have major cardiovascular disease within 6 months before screening, which includes, but not limited to Severe heart disease (heart failure (NYHA class 3 and 4), acute coronary artery disease (unstable angina, acute myocardial infarction), clinically significant ventricular tachycardia, atrial fibrillation, atrial flutter, or other clinically significant arrhythmia and peripheral vascular diseases confirmed by the investigator Hypertrophic obstructive cardiomyopathy, clinically significant heart valve disease or aortic disease
   * Patients who are considered inappropriate to participate in the study because they have uncontrolled disease and have a comorbid disease that requires treatment by the investigator's judgement (e.g., blood coagulation disorder, bleeding disorder or bleeding diatheses, pulmonary function decline, decline in renal function, hypotension, hypertension, hepatitis, liver cirrhosis, etc)
   * Patients who have major mental illness (e.g., depression, bipolar disorder, etc.) or a history of drug/alcohol abuse
2. If the following therapy has been administered or received, or when the need for administration is expected

   * The following therapies within 12 weeks before the baseline that may have a significant effect on the results of the study Palifermin Oral low-level laser therapy Oral cryotherapy Glutamine (parenteral, IV supplement of protein amino acids containing glutamic acid, not glutamine supplements, are permitted)
   * Vaccination of yellow fever vaccine or other live attenuated vaccine within 4 weeks before the baseline
   * Anti-cancer or radiation therapy* within 3 weeks before the baseline (However, the use of Anti-cancer drugs for hematopoietic stem cell collection is permitted and subjects who have been irradiated with head and neck within the last 2 years are excluded.) (*Radio(chemo)therapy, chemotherapy, targeted therapy (small molecule drugs, monoclonal antibodies), cancer immunotherapy (biological drugs), or hormone therapy, etc.)
   * The following drugs that may affect the metabolism of IP from within 7 days before the baseline to the end of treatment (EOT) period Strong CYP3A4 inhibitors: boceprevir, citrus x paradisi, clarithromycin, cobicistat, conivaptan, delavirdine, diltiazem, idelalisib, indinavir, itraconazole, ketoconazole, mibefradil, miconazole, nefazodone, nelfinavir, posaconazole, lopinavir/ritonavir, saquinavir, telaprevir, telithromycin, tipranavir, troleandomycin, voriconazole Strong CYP3A4 inducers: avasimibe, carbamazepine, enzalutamide, fosphenytoin, hypericum perforatum, lumacaftor, methylphenobarbital, mitotane, phenobarbital, phenobarbital quinine, primidone, rifabutin, rifampicin, rifapentine OATP inhibitors: cyclosporin A, cyclosporine, estradiol-17β-glucuronide, estrone-3-sulfate, rifampicin, rifamycin SV, lopinavir/ritonavir
3. Pregnant and lactating women or women or childbearing potential and men who have a pregnancy plan up to 30 days after the end of the IP administration or who do not intend to use appropriate contraception: ① Hormonal contraceptives, ② Implantation of an intrauterine device or intrauterine system, ③ Double blocking method with spermicide (both male condom and closed cap (contraceptive diaphragm or neck cap) are used), ④ Infertility procedures (e.g., vasectomy, bilateral tubal ligation, etc.)
4. Patients who participated in other clinical trials within 30 days from the start of IP administration and received other study drug (or medical devices)
5. Patient who are judged to be difficult to participate in the study according to the opinions of investigators

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
The incidence of Severe Oral Mucositis(SOM). | up to 14 days after the end of therapy( or discharge if hospitalization extension is necessary)
  OM is evaluated using the World Health Organization (WHO) OM grading scale that uses a scale of 0 to 4.
  SOM is defined as a WHO score of greater than or equal to 3.
  OM grading scale
  Grade 0 = Normal
  Grade 1 = Erythema and Soreness
  Grade 2 = Ulceration but can eat solid foods
  Grade 3 = Ulceration,diet limited to liquid (due to mucositis)
  Grade 4 = Ulceration of severity that patient requires parenteral feeding (due to mucositis)

SECONDARY OUTCOMES:
The incidence of oral mucositis by WHO OM grading scale | up to 14 days after the end of therapy( or discharge if hospitalization extension is necessary)
  ① Grade 1 or higher, ② Grade 2 or higher, ③ Grade 4 or higher
  OM grading scale
  Grade 0 = Normal
  Grade 1 = Erythema and Soreness
  Grade 2 = Ulceration but can eat solid foods
  Grade 3 = Ulceration,diet limited to liquid (due to mucositis)
  Grade 4 = Ulceration of severity that patient requires parenteral feeding (due to mucositis)
The incidence of oral mucositis based on the maximum severity by WHO OM grading scale | up to 14 days after the end of therapy( or discharge if hospitalization extension is necessary)
  ① Grade 1 ② Grade 2 ③ Grade 3 ④ Grade 4
  OM grading scale
  Grade 0 = Normal
  Grade 1 = Erythema and Soreness
  Grade 2 = Ulceration but can eat solid foods
  Grade 3 = Ulceration,diet limited to liquid (due to mucositis)
  Grade 4 = Ulceration of severity that patient requires parenteral feeding (due to mucositis)
The average grade of oral mucositis by WHO OM grading scale | Each 1, 5, 7, 14, 21 and 28 day after the end of therapy
  The average grade of each point
  OM grading scale
  Grade 0 = Normal
  Grade 1 = Erythema and Soreness
  Grade 2 = Ulceration but can eat solid foods
  Grade 3 = Ulceration,diet limited to liquid (due to mucositis)
  Grade 4 = Ulceration of severity that patient requires parenteral feeding (due to mucositis)
The duration of oral mucositis by WHO OM grading scale | up to 14 days after the end of therapy( or discharge if hospitalization extension is necessary)
  ① Grade 2 or higher, ② Grade 3 or higher, ③ Grade 4 or higher
  OM grading scale
  Grade 0 = Normal
  Grade 1 = Erythema and Soreness
  Grade 2 = Ulceration but can eat solid foods
  Grade 3 = Ulceration,diet limited to liquid (due to mucositis)
  Grade 4 = Ulceration of severity that patient requires parenteral feeding (due to mucositis)
The incidence of oral mucositis by NCI-CTCAE v5.0 criteria | up to 14 days after the end of therapy( or discharge if hospitalization extension is necessary)
  ① Grade 1 or higher, ② Grade 2 or higher, ③ Grade 3 or higher, ④ Grade 4 or higher
  Grade 0 = Normal
  Grade 1 = Asymptomatic or mild symptoms; intervention not indicated
  Grade 2 = Moderate pain or ulcer that does not interfere with oral intake; modified diet indicated
  Grade 3 = Severe pain; interfering with oral intake
  Grade 4 = Life-threatening consequences; urgent intervention indicated
  Grade 5 = Death
The average grade of oral mucositis by NCI-CTCAE v5.0 criteria | Each 1, 5, 7, 14, 21 and 28 day after the end of therapy
  The average grade of each point
  Grade 0 = Normal
  Grade 1 = Asymptomatic or mild symptoms; intervention not indicated
  Grade 2 = Moderate pain or ulcer that does not interfere with oral intake; modified diet indicated
  Grade 3 = Severe pain; interfering with oral intake
  Grade 4 = Life-threatening consequences; urgent intervention indicated
  Grade 5 = Death
The mean area under curve(AUC) of score for each question in oral mucositis daily questionnaire(OMDQ) | up to 14 days after the end of therapy( or discharge if hospitalization extension is necessary)
  Q1: General health condition scale: 0(worst possible) to 10(perfect health)
  Q2: Mouth and throat pain: 0(no soreness) to 4(extreme soreness)
  Q3: Salvia swallowing, drinking water, eat rice, speaking ans sleeping: 0(no soreness) to 4(extreme soreness)
  Q4: General mouth and throat pain: 0(no soreness) to 10(worst possible)
The proportion of using opioid analgesics | From the baseline to 14 days after the end of therapy( or discharge if hospitalization extension is necessary)
  The proportion of patients who used opioid analgesics up to 14 days after the end of therapy.
Total cumulative dose of opioid analgesics | From the baseline to 14 days after the end of therapy( or discharge if hospitalization extension is necessary)
  It will be calculated as morphine equivalents dose

OTHER OUTCOMES:
Adverse Events(AEs) | From baseline to 28 day after discharge
  The number and incidence rate of AEs will be investigated.
Auto hematopoietic stem cell engraftment | From auto-HSCT to 28 day
  * achievement of ANC > 0.5x10^9/L for three consecutive days
  * achievement of peripheral platelet > 20 X 10^9/L for three consecutive days

CONTACTS AND LOCATIONS:
Overall Officials: Seok-Goo Cho, MD, PhD, Principal Investigator — Seoul St. Mary's Hospital
Locations (2):
- South Korea (2):
  - Seoul ST. Mary's Hospital, Seoul
  - Yeouido ST. Mary's Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No